CLINICAL TRIAL: NCT01366313
Title: The Median Effective Dose (ED50) of Paracetamol and Morphine for Postoperative Patients: A Study of Interaction.
Brief Title: The Median Effective Dose (ED50) of Paracetamol and Morphine : A Study of Interaction Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procare Riaya Hospital (Other)
Responsible Party: Principal Investigator, Ahed ZEIDAN, MD, Procare Riaya Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRH 02
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2011-01

CONDITIONS: Postoperative Pain
Keywords: paracetamol; morphine; median effective dose; pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Acetaminophen; Morphine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Paracetamol (Experimental): initial doses was 1.5g g, with dose adjustment intervals of 0.5g . with maximum dose 2.5 g as an only starting dose / 24 h
  Interventions: Drug: Paracetamol
- Morphine (Experimental): Initial doses of morphine was 5mg, with dose adjustment intervals of 1 mg .
  Interventions: Drug: Morphine
- Paracetamol-morphine (Experimental): The initial doses of paracetamol and morphine were 1.5g and 3mg, respectively in the paracetamol-morphine combination group with dose adjustment intervals of 0.25g for paracetamol and 0.5mg for morphine.
  Interventions: Drug: Paracetamol- Morphine

INTERVENTIONS:
Drug: Paracetamol — initial doses was 1.5g, with dose adjustment intervals of 0.5g . with maximum dose 2.5 g as an only starting dose / 24 h
  Other Names: Perfalgan
  Arms: Paracetamol
Drug: Morphine — Initial of morphine was 5mg, with dose adjustment intervals 1 mg .
  Other Names: Morphine sulfate
  Arms: Morphine
Drug: Paracetamol- Morphine — The initial doses of paracetamol and morphine were 1.5g and 3mg, respectively in the paracetamol-morphine combination group with dose adjustment intervals of 0.25g for paracetamol and 0.5mg for morphine.
  Other Names: Perfalgan-Morphine
  Arms: Paracetamol-morphine

SUMMARY:
The aim of our study is to define the median effective analgesic doses (ED50) of paracetamol, morphine, and their combination and determination the nature of their interaction administered IV for postoperative pain after moderate painful surgery using up-and-down and isobolographic methods.

DETAILED DESCRIPTION:
Ninety patients scheduled to undergo moderately painful surgery were included in one of three groups. Determination of median effective (ED50) doses was performed by the Dixon and Mood up-and-down method. Initial doses were 1.5g and 5mg, with dose adjustment intervals of 0.5g and 1 mg, in the paracetamol and morphine groups, respectively. The initial doses of paracetamol and morphine were 1.5g and 3mg, respectively in the paracetamol-morphine combination group with dose adjustment intervals of 0.25g for paracetamol and 0.5mg for morphine. Analgesic efficacy was defined as a decrease to less than 3 on a 0-10 numeric pain scale, 45 min after the beginning of drug administration. Isobolographic analysis was used to define the nature of their interaction.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status І or ІІ
2. Moderately painful surgery patients
3. postoperative pain more than 3 on a numerical pain score (NPS) -

Exclusion Criteria:

1. contraindication to the use of paracetamol and morphine
2. Pregnancy
3. age younger than 18 yr
4. patient weight less 65kg
5. intra-operative regional anesthesia,
6. intra-operative administration of analgesics other than fentanyl,
7. postoperative pain less than 3 on a numerical pain score (NPS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
ED50s of Paracetamol, morphine and their combination | participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  the aim of our study is to define the median effective analgesic doses (ED50s) of paracetamol, morphine, and their combination to determine the nature of their interaction administered IV for postoperative moderately painful surgery using the Dixon and Mood up-and-down method and isobolographic analysis.

SECONDARY OUTCOMES:
Paracetamol-Morphine interaction nature | participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  the aim of our study is to define the median effective analgesic doses (ED50s) of paracetamol, morphine, and their combination to determine the nature of their interaction administered IV for postoperative moderately painful surgery using the Dixon and Mood up-and-down method and isobolographic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: AHED ZEIDAN, MD, Study Chair — Procare Riaya Hospital
Locations (1):
- Procare Riaya Hospital, Khobar, Estern, Saudi Arabia

REFERENCES:
- [Derived] Zeidan A, Mazoit JX, Ali Abdullah M, Maaliki H, Ghattas T, Saifan A. Median effective dose (ED(5)(0)) of paracetamol and morphine for postoperative pain: a study of interaction. Br J Anaesth. 2014 Jan;112(1):118-23. doi: 10.1093/bja/aet306. Epub 2013 Oct 24. PMID 24157897